CLINICAL TRIAL: NCT02146976
Title: Postoperative Sleep Quality of Patients Anesthesia With Propofol or Sevoflurane Undergoing Thyroidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20140522
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Sleep Quality
Keywords: postoperative; sleep quality; propofol; sevoflurane
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Experimental): introvenious infusion of propofol
  Interventions: Drug: propofol
- Inhaled anaesthetic (Sevoflurane) (Experimental): sevoflurane (1.0-1.3% Minimum Alveolar Concentration)
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — introvenious infusion of propofol
  Arms: Propofol
Drug: sevoflurane — sevoflurane (1.0-1.3 Minimum Alveolar Concentration)
  Arms: Inhaled anaesthetic (Sevoflurane)

SUMMARY:
The investigators designed a study to determine whether Propofol or Sevoflurane would provide same postoperative sleep quality in patients undergoing thyroidectomy.

DETAILED DESCRIPTION:
The investigators designed a study to determine whether Propofol or Sevoflurane would provide same postoperative sleep quality in patients undergoing thyroidectomy.The bispectral index score (BIS) was monitored during the operation and the first postoperative night.

ELIGIBILITY:
Inclusion Criteria:

* Participants were deemed eligible if they were candidates for general anesthesia undergoing thyroidectomy

Exclusion Criteria:

* Patients were excluded if they had a body mass index exceeding 30 kg/m2, had a Pittsburgh Sleep Quality Index global scores higher than 6, had an anesthesia time longer than 4 hours, had a history of cardiovascular, neurological, or psychiatric disease, had cervical lymph node metastasis, were treated with sedative and analgesics during the postoperative BIS-Vista monitoring period, were allergic to drugs used in the study, or had been diagnosed with Graves' disease or hyperthyroidism or hypothyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The Change of postoperative sleep quality | preoperation, first postoperative night
  The primary outcome was the postoperative sleep quality, which was measured by the BIS-Vista monitor on the first night after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,Ph.D., Study Chair — the Anesthesiology Department
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided